CLINICAL TRIAL: NCT01663155
Title: A Clinical Trial to Develop Chest Imaging, Breath, and Biomarkers in a Screening Trial
Brief Title: Chest Imaging, Breath, and Biomarkers in a Screening Trial
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Moulay Meziane, MD, Principal Investigator, The Cleveland Clinic
Other Study IDs: 07-455; State of Ohio grant (Other Grant/Funding Number: 06-055); 06-055 (Other Grant/Funding Number: State of Ohio)
Record Dates: First submitted 2008-11-10; First posted 2012-08-13 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Lung Cancer
Keywords: lung cancer; chest x-ray; CT scan; computer aided detection (CAD); screening; smokers
MeSH Terms: conditions — Lung Neoplasms | interventions — Diagnostic Imaging; Diagnosis, Computer-Assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood draw includes 2 10 mL red top tubes for serum retrieval, and 2 7 mL EDTA tubes for plasma and buffy coat retrieval
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- all enrolled subjects: Intervention is chest x-ray and CT scan. The chest x-ray image is read first without computer aided detection (CAD) and then a second time with computer aided detection (CAD) the CT scan is read by one reader. Subjects are asked to contribute breath and blood samples.
  Interventions: Device: chest x-ray with or without CAD, lose dose CT scan

INTERVENTIONS:
Device: chest x-ray with or without CAD, lose dose CT scan — PA view, low dose CT scan
  Other Names: CAD; computer aided detection

SUMMARY:
The investigators would like to see if lung cancer screening with chest x-rays,computer aided detection (CAD)and a lose dose CT scan can detect lung cancer in early stages when it is more responsive to treatment. The investigators would also like to see if early detection will reduce the incidence of symptomatic advanced lung cancer compared to no screening in former and current smokers with or without a family history of lung cancer who are 40-75 years old.

DETAILED DESCRIPTION:
The fight against lung cancer is waged on three major fronts: prevention, detection and treatment. Our goal is to determine if chest x-rays,computer aided detection (CAD)and a CT scan can detect disease earlier when treatment is more effective. If we improve the detection of disease, we will see if screening reduces the incidence of symptomatic advanced lung cancer relative to no screening in people at high risk to develop lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* ages 40-75 years
* If ages 40-59, then one of the following criteria needs to be met:

  * Current or ex-smoker with >25 pack years and a family history of lung cancer(parent or sibling) OR
  * current or ex-smoker with > 25 pack years and COPD OR
  * current or ex-smoker with a > 35 pack year history
* If ages 60-75, then one of the following additional criteria needs to be met:

  * Current or ex-smoker with >25 pack years and a family history of lung cancer (parent or sibling) OR
  * Current or ex-smoker with >25 pack years and COPD OR
  * Current or ex-smoker with a >30 pack year history
* Subject is able to return to Cleveland Clinic for annual follow-up screening
* Subject is willing to sign a medical release form

Exclusion Criteria:

* Current health requires oxygen
* Have had a chest x-ray or CT of the chest within the last 6 months
* Previous pneumonectomy
* Lobectomy of the lung within the last 5 years
* Diagnosed malignancy within the last 5 years, excluding non-melanoma skin cancer, carcinoma in situ of the cervix and localized prostate cancer
* A medical condition that would prevent treatment for lung cancer
* Within the last 6 weeks, one of the following has occured:

  * A new cough or chronic cough that has gotten worse
  * Either new shortness of breath, or any worsening of shortness of breath
  * A cough producing blood
  * Constant chest pain
  * Respiratory infection, pneumonia, or cold
  * Unintentional and unexplained weight loss greater than 5% of total body weight

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care physicians or any other physician may refer potential candidates. Additionally, subjects may see marketing materials and contact the research team directly. There is no restriction to the area of residence of subjects.
Sampling Method: Probability Sample
Enrollment: 1424 (Actual)
Dates: Start 2008-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The sensitivities of chest x-ray with CAD and chest CT | One year after scan
  The false positive rates of chest x-ray with CAD and chest CT will be compared. The analysis will be based on the study subjects from this prospective study who test positive with chest x-ray and/or CT and who are determined not to have lung cancer during the follow-up period.

SECONDARY OUTCOMES:
Disease-specific mortality between screening with chest x-ray and CAD versus no screening | One year after scan
  Mortality rate in screening x-ray vs CAD
All-cause mortality rate between screening with chest x-ray and CAD versus no screening | One year after scan
  All cause mortality rate
Length of time between randomization and the incidence of symptomatic advanced lung cancer for screened subjects versus controls | One year after scan
  Time between randomization and symptom
Does lung cancer screening with chest x-rays and computer aided detection (CAD) reduce the incidence of symptomatic advanced lung cancer in a high risk population | One year after scan
  Cancer detection rate between chest x-ray and CAD
The quality of life between screening with chest x-ray and CAD versus no screening. | One year after scan
  Quality of life between the chest x-ray group and the CAD group

CONTACTS AND LOCATIONS:
Overall Officials: Micheal Phillips, M.D., Study Chair — The Cleveland Clinic; Moulay Meziane, MD, Principal Investigator — Chair of Thoracic Imaging
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Mazzone PJ, Obuchowski N, Fu AZ, Phillips M, Meziane M. Quality of life and healthcare use in a randomized controlled lung cancer screening study. Ann Am Thorac Soc. 2013 Aug;10(4):324-9. doi: 10.1513/AnnalsATS.201301-007OC. PMID 23952850
- [Derived] Mazzone PJ, Obuchowski N, Phillips M, Risius B, Bazerbashi B, Meziane M. Lung cancer screening with computer aided detection chest radiography: design and results of a randomized, controlled trial. PLoS One. 2013;8(3):e59650. doi: 10.1371/journal.pone.0059650. Epub 2013 Mar 20. PMID 23527241